CLINICAL TRIAL: NCT02172287
Title: A Multiple Dose Comparison of Tiotropium Inhalation Capsules, Salmeterol Inhalation Aerosol and Placebo in a Six-Month, Double-Blind, Double-Dummy, Safety and Efficacy Study in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Multiple Dose Comparison of Tiotropium Inhalation Capsules, Salmeterol Inhalation Aerosol and Placebo in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.130
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate

ARMS (3):
- Tiotropium (Ba679 BR) (Experimental): Tiotropium capsule once daily by oral inhalation
  Interventions: Drug: Tiotropium (Ba679 BR); Drug: Placebo (for Salmeterol)
- Salmeterol (Active Comparator): Salmeterol inhalation aerosol twice daily
  Interventions: Drug: Salmeterol; Drug: Placebo (for Tiotropium )
- Placebo (Placebo Comparator): * Tiotropium (Ba679 BR)- placebo one capsule once daily by inhalation
  * Salmeterol- placebo, inhalation aerosol twice daily
  Interventions: Drug: Placebo (for Tiotropium ); Drug: Placebo (for Salmeterol)

INTERVENTIONS:
Drug: Tiotropium (Ba679 BR) — One capsule once daily by oral inhalation
  Arms: Tiotropium (Ba679 BR)
Drug: Salmeterol — Inhalation aerosol twice daily
  Arms: Salmeterol
Drug: Placebo (for Tiotropium ) — Placebo for Tiotropium delivered by inhalation capsule
  Arms: Placebo; Salmeterol
Drug: Placebo (for Salmeterol) — Placebo for Salmeterol delivered by inhalation aerosol
  Arms: Placebo; Tiotropium (Ba679 BR)

SUMMARY:
To compare the long -term (six month) bronchodilator efficacy and safety of tiotropium inhalation capsules, salmeterol inhalation aerosol and placebo in patients with COPD. A secondary objective of this study was to compare the impact of tiotropium and salmeterol on humanistic and economic health outcomes, such as quality of life, patient preference and Health Resource Utilisation in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years.
2. A diagnosis of relatively stable, moderate to severe COPD with:
3. Screening FEV1 ≤ 60% of predicted normal value (calculated according to European Community for Coal and Steel (ECCS criteria R94- R1408) and screening FEV1 ⁄ FVC ≤ 70%).
4. Smoking history ≥ 10 pack-years (a pack-year is 20 cigarettes per day for one year or equivalent).
5. Ability to be trained in the proper use of the HandiHaler® device and Mahler Dyspnoea Index (MDI).
6. Ability to perform all study related tests including the Shuttle Walking Test, acceptable pulmonary function tests, including Peak Expiratory Flow Rate (PEFR) measurements, and maintenance of daily diary card records.
7. Ability to give written informed consent in accordance with Good Clinical Practice (GCP) and local regulations.

Exclusion Criteria:

1. Clinically significant diseases other than COPD. A clinically significant disease is defined as one which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion, will be excluded.
3. All patients with a serum glutamic oxaloacetic transaminase (SGOT) > 80 IU/L, serum glutamic pyruvic transaminase (SGPT) > 80 IU/L, bilirubin > 2.0 mg/dL or creatinine > 2.0 mg/dL will be excluded regardless of clinical condition. Repeat laboratory evaluation should have not been conducted in these patients.
4. A recent history (i.e., one year or less) of myocardial infarction.
5. Any cardiac arrhythmia requiring drug therapy or hospitalisation for heart failure within the past three years.
6. Inability to abstain from regular daytime use of oxygen therapy for more than 1 hour per day.
7. Known active tuberculosis.
8. History of cancer within the last five years (excluding basal cell carcinoma).
9. History of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
10. Patients who have undergone thoracotomy with pulmonary resection.
11. Any upper respiratory infection in the past six weeks prior to the screening visit or during the run-in period.
12. Current participation in a pulmonary rehabilitation programme or completion of a pulmonary rehabilitation programme in the six week prior to the screening visit.
13. Known hypersensitivity to anticholinergic drugs, salmeterol, or any of the components of the lactose powder capsule or MDI delivery systems.
14. Known symptomatic prostatic hypertrophy or bladder neck obstruction.
15. Patients with known narrow-angle glaucoma.
16. Current treatment with cromolyn sodium or nedocromil sodium.
17. Current treatment with antihistamines (H1 receptor antagonists).
18. Oral corticosteroids medication at unstable doses (i.e. less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg prednisolone per day or 20 mg every other day.
19. Current use of β-blocker medication.
20. Current treatment with monoamine oxidase inhibitors of tricyclic and antidepressants.
21. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception.
22. Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count ≥ 600 mm3. A repeat eosinophil count was not permitted.
23. History of and/or active significant alcohol or drug abuse.
24. Concomitant or recent use of an investigational drug within one month or six half lives (whichever is greater) prior to the screening visit.
25. Changes in the pulmonary therapeutic plan within the six weeks prior to the screening visit.
26. Inability to comply with the medication restrictions specified in Section 4.2 of the trial protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 1999-02; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in trough Forced expiratory volume in one second (FEV1) response | baseline, up to day 169
Change from baseline in Mahler Transitional Dyspnoea Index (TDI) | baseline, up to day 169

SECONDARY OUTCOMES:
Average Forced Expiratory Volume (FEV1) response on each test-day | 60 and 10 minutes before in-clinic dosing and at 30 minutes and 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post-dose on day 1, 15, 57, 113 and 169
Peak Forced Expiratory Volume (FEV1) response on each test-day | 60 and 10 minutes before in-clinic dosing and at 30 minutes and 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post-dose on day 1, 15, 57, 113 and 169
Trough Forced Vital Capacity (FVC) on each test day | 60 and 10 minutes before in-clinic dosing and at 30 minutes and 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post-dose on day 1, 15, 57, 113 and 169
Average Forced Vital Capacity (FVC) on each test day | 60 and 10 minutes before in-clinic dosing and at 30 minutes and 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post-dose on day 1, 15, 57, 113 and 169
Peak of Forced Vital Capacity (FVC) on each test day | 60 and 10 minutes before in-clinic dosing and at 30 minutes and 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post-dose on day 1, 15, 57, 113 and 169
Individual FEV1 measurements at each time point | 60 and 10 minutes before in-clinic dosing and at 30 minutes and 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post-dose on day 1, 15, 57, 113 and 169
Individual FVC measurements at each time point | 60 and 10 minutes before in-clinic dosing and at 30 minutes and 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post-dose on day 1, 15, 57, 113 and 169
Peak Expiratory Flow Rate (PEFR) measured by the patients at home | twice daily for 29 weeks
Change from baseline in Physicians global evaluation | baseline, day 15, 57, 113, 169 and 190
Change from baseline in Chronic Obstructive Pulmonary Disease (COPD) symptom score | baseline, day 15, 57, 113, 169 and 190
Amount of rescue medication (salbutamol) therapy used during the treatment period | up to day 169
Number and length of exacerbations of COPD during the treatment period | up to day 169
Number and length of hospitalisations for respiratory disease during the treatment period | up to day 169
Change from baseline in Quality of Life measures using St. George's Respiratory Questionnaire (SGRQ) | baseline, day 57, 113, 169 and 190
Health resource utilisation beyond the study protocol | up to day 190
Change in Patient preference measures (satisfaction with COPD medication) | baseline, day 169
Change from baseline in Shuttle walking tests | baseline, day 57, 113, 169 and 190
Change from baseline in Borg dyspnea score | baseline, day 57, 113, 169 and 190
Number of patients with adverse events | up to day 190
Change from baseline Pulse rate and blood pressure | baseline, day 57, 113 and 169
Change from baseline in laboratory tests | baseline, day 169
Change from baseline in ECG | baseline, day 169